CLINICAL TRIAL: NCT02048397
Title: A Pilot Study of Pulmonary Rehabilitation Program (PRP) Versus PRP Plus Nutritional Supplementation in Patients With Bronchiectasis: a Randomized Controlled Trial
Brief Title: Pulmonary Rehabilitation Program (PRP) Versus PRP Plus Nutritional Supplementation in Patients With Bronchiectasis
Acronym: FIM-BRO-2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIM-BRO-2013-01
Record Dates: First submitted 2014-01-15; First posted 2014-01-29 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2013-08

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis.
MeSH Terms: conditions — Bronchiectasis | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary Rehabilitation (PRP) (Other): Pulmonary Rehabilitation (PRP)
  Interventions: Other: Pulmonary Rehabilitation
- Pulmonary Rehabilitation plus oral nutritional supplement (Other): Hyperproteic oral nutritional supplement enriched with beta-hydroxy-beta-methylbutyrate (HMB)
  Interventions: Dietary Supplement: Hyperproteic oral nutritional supplement enriched with beta-hydroxy-beta-methylbutyrate

INTERVENTIONS:
Other: Pulmonary Rehabilitation
  Arms: Pulmonary Rehabilitation (PRP)
Dietary Supplement: Hyperproteic oral nutritional supplement enriched with beta-hydroxy-beta-methylbutyrate
  Arms: Pulmonary Rehabilitation plus oral nutritional supplement

SUMMARY:
The effect of Pulmonary Rehabilitation in patients with bronchiectasis (BC) is not sufficiently studied. The aim of this study is to assess the clinical and biological response of a Pulmonary Rehabilitation Program (PRP) for 12 weeks in BC vs PRP plus hyperproteic oral nutritional supplement enriched with beta-hydroxy-beta-methylbutyrate (HMB).

Methods: single center randomized controlled trial, parallel treatment design: Participants will be randomized assigned either will receive (n=14) PRP for 60 minutes, two supervised sessions per week in the hospital and one unsupervised session at home vs PRP (n=14) plus ONS (one can per day).

Outcome assessments will be performed at baseline, 12 weeks and 24 weeks:

1.- effort capacity –cardiopulmonary exercise test-, 2.- body composition (anthropometry, lean body mass by dual energy X-ray absorptiometry and bioimpedance, phase angle), 3.- peripheral muscle strength (dynamometry and respiratory -PEM (maximum expiratory pressure)and PIM (minimum expiratory pressure)-), 4.- spirometry, 5.- respiratory symptoms (bronchorrhea, dyspnoea, exacerbations),6.- level of physical activity (IPAQ questionnaire plus objective physical activity (WGT3X)), 7.- quality of life (QOL-B-Spain) , 8.-psychological symptoms (HASD) and 9.- biological markers of inflammation (leptin, adiponectin, interleukin-6, tumor necrosis factor-alpha, ultrasensitive C-reactive protein, GPR55 (G protein-coupled receptor 55) RNAm (messenger ribonucleic acid) expression in white blood cells) and oxidation (total antioxidant capacity, superoxide dismutase activity, 8-iso-prostaglandin F2a, Thiobarbituric acid reactive substances).

ELIGIBILITY:
Inclusion Criteria:

* Patients ages from 18-80 (both included)
* Patients with bronchiectasis, not cystic fibrosis bronchiectasis.
* Bronchiectasis diagnosed by high resolution computed tomography (HRCT). of the chest
* Patients followed in Bronchiectasis and Cystic Fibrosis Units in the Hospital.
* BMI > 18.5 in patients under 65 years old, and > 20kg/m2 in patients over this age.
* Ambulatory patients.

Exclusion Criteria:

* Use of oral corticoids.
* Respiratory exacerbation. If a patient had a respiratory exacerbation or a recent hospital admission, their participation will be postponed for at least 60 days til any acute disease is resolved.
* Prior oral or parenteral supplements intake.
* Traumatological, neurological or cardiovascular diseases that prevent patients from performing the training.
* Life threatening hemoptysis in the past year.
* Patients with cancer, major surgery in the previous three months, participating in another study, patients who are pregnant or may become pregnant, patients with acute intestinal disease, acute heart failure, severe hepatic failure or dialysis.
* Gastrectomy, gastroparesis or other alterations of gastric emptying.
* Enteral tube feeding, galactosemia, Fructosemia.
* Allergy or known sensitivity to any ingredient of the enteral formula.
* Cystic fibrosis.
* Included in active list for transplantation.
* Drug or alcohol abuse.
* No informed consent signed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in oxygen uptake at peak exercise (VO2max) in cardiopulmonary exercise test (Before and after Rehabilitation-at 3 and 6 months) | 3rd and 6th month visits

SECONDARY OUTCOMES:
Body composition | 3rd and 6th month visits
  Anthropometry, lean body mass by dual energy X-ray absorptiometry and bioimpedance.

OTHER OUTCOMES:
Peripheral muscle strength | 3rd and 6th month visits
  Dynamometry
Change from baseline in respiratory symptoms (bronchorrhea, dyspnea, exacerbations) at 6 months. | 3rd and 6th month visits
Level of physical activity | 3rd and 6th month visits
  IPAQ questionnaire plus objective physical activity
Quality of life | 3rd and 6th month visits
  QOL-B-Spain
biological markers of Biological markers of inflammation and oxidation | 3rd and 6th month visits

CONTACTS AND LOCATIONS:
Overall Officials: GABRIEL OLVEIRA, MD, PhD, Principal Investigator — Andaluz Health Service
Locations (1):
- Gabriel Olveira, Málaga, Malaga, Spain

REFERENCES:
- [Background] Clin Nutr. 2015 Oct 19. pii: S0261-5614(15)00255-1. doi: 10.1016/j.clnu.2015.10.001. [Epub ahead of print]
- [Derived] Dona E, Olveira C, Palenque FJ, Porras N, Dorado A, Martin-Valero R, Godoy AM, Espildora F, Olveira G. Pulmonary Rehabilitation Only Versus With Nutritional Supplementation in Patients With Bronchiectasis: A RANDOMIZED CONTROLLED TRIAL. J Cardiopulm Rehabil Prev. 2018 Nov;38(6):411-418. doi: 10.1097/HCR.0000000000000341. PMID 29952809
- [Derived] Dona E, Olveira C, Palenque FJ, Porras N, Dorado A, Martin-Valero R, Godoy AM, Espildora F, Contreras V, Olveira G. Body Composition Measurement in Bronchiectasis: Comparison between Bioelectrical Impedance Analysis, Skinfold Thickness Measurement, and Dual-Energy X-ray Absorptiometry before and after Pulmonary Rehabilitation. J Acad Nutr Diet. 2018 Aug;118(8):1464-1473. doi: 10.1016/j.jand.2018.01.013. Epub 2018 Apr 12. PMID 29656933
- [Derived] Olveira G, Olveira C, Dona E, Palenque FJ, Porras N, Dorado A, Godoy AM, Rubio-Martinez E, Rojo-Martinez G, Martin-Valero R. Oral supplement enriched in HMB combined with pulmonary rehabilitation improves body composition and health related quality of life in patients with bronchiectasis (Prospective, Randomised Study). Clin Nutr. 2016 Oct;35(5):1015-22. doi: 10.1016/j.clnu.2015.10.001. Epub 2015 Oct 19. PMID 26522923